CLINICAL TRIAL: NCT01396824
Title: Nutrition Status and Body Composition in Ambulatory Patients With Heart Failure and Its Prognostic Significance (PLiegues en Insuficiencia Cardiaca-PLICA).
Brief Title: Nutritional Status and Prognosis in Heart Failure.
Acronym: PLICA
Status: Completed | Type: Observational
Sponsor: Germans Trias i Pujol Hospital (Other)
Responsible Party: Principal Investigator, Antoni Bayés Genís, Chief of the Cardiology Service, Germans Trias i Pujol Hospital
Other Study IDs: ICREC-2011-01
Record Dates: First submitted 2011-07-18; First posted 2011-07-19 (Estimated); Last update posted 2016-06-02 (Estimated); Status verified 2016-06

CONDITIONS: Heart Failure
Keywords: Malnutrition; Undernutrition; Nutrition Assessment; Nutritional Assessment; Nutritional Index; Prognostic Nutritional Index; Prognostic Nutritional Index (PNI); Nutritional Status; Prognosis; Heart Failure; Cardiovascular Diseases; Body Composition; Body Weights and Measures
MeSH Terms: conditions — Heart Failure; Malnutrition; Cardiovascular Diseases; Body Weight

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Heart failure: Heart failure patients attending a HF clinic with depressed LVEF (< 45%) or ≥ 1 hospital admission due to HF decompensation.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
The purpose of this study is to determine whether nutritional status or body composition influences the prognosis of heart failure patients.

DETAILED DESCRIPTION:
Despite obesity is a cardiovascular risk factor, numerous studies have identified a better prognosis in overweight and obese heart failure (HF) patients. This paradox has been named "the obesity paradox". However, this paradox has been criticized because the parameter used to classify obesity, the body mass index (BMI), has several limitations. Obesity is defined as an abnormal or excessive fat accumulation, and BMI does not always reflect real body fat.

What is more, patients with HF can have their body composition altered with hyperhydration or undernourishment. A pilot study proved that BMI does not indicate true nutritional status in HF. Thus, a further assessment of body composition of HF patients, analyzing the nutritional status rather BMI, could shed light on the obesity paradox. The aim of this study was to assess the nutritional status of a cohort of HF patients, its correspondence with BMI, and its significance in terms of survival.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of heart failure according to the European Guidelines of Heart Failure.
* Depressed LVEF (< 45%) or ≥ 1 hospital admission due to HF decompensation
* Outpatients > 18 years of age, male or female, capable of giving an informed consent.

Exclusion Criteria:

* Severe co-morbidity associated with a reduction in life expectancy of less than 1 year.
* Myopathy or other diseases that could cause significant sarcopenia beyond HF.
* Non-controlled hyperthyroidism

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive heart failure patients attending the HF clinic of a university hospital.
Sampling Method: Probability Sample
Enrollment: 214 (Actual)
Dates: Start 2011-06; Primary Completion 2013-07 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
All cause mortality | 3 years

SECONDARY OUTCOMES:
Cardiac mortality and non-cardiac mortality | 3 years
Heart failure hospitalizations | 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- Germans Trias Research Institute; Germans Trias University Hospital, Badalona, Barcelona, Spain

REFERENCES:
- [Background] Lavie CJ, Milani RV, Artham SM, Patel DA, Ventura HO. The obesity paradox, weight loss, and coronary disease. Am J Med. 2009 Dec;122(12):1106-14. doi: 10.1016/j.amjmed.2009.06.006. Epub 2009 Aug 13. PMID 19682667
- [Background] Curtis JP, Selter JG, Wang Y, Rathore SS, Jovin IS, Jadbabaie F, Kosiborod M, Portnay EL, Sokol SI, Bader F, Krumholz HM. The obesity paradox: body mass index and outcomes in patients with heart failure. Arch Intern Med. 2005 Jan 10;165(1):55-61. doi: 10.1001/archinte.165.1.55. PMID 15642875
- [Background] Lavie CJ, Milani RV, Ventura HO, Romero-Corral A. Body composition and heart failure prevalence and prognosis: getting to the fat of the matter in the "obesity paradox". Mayo Clin Proc. 2010 Jul;85(7):605-8. doi: 10.4065/mcp.2010.0333. No abstract available. PMID 20592168
- [Background] Kalantar-Zadeh K, Block G, Horwich T, Fonarow GC. Reverse epidemiology of conventional cardiovascular risk factors in patients with chronic heart failure. J Am Coll Cardiol. 2004 Apr 21;43(8):1439-44. doi: 10.1016/j.jacc.2003.11.039. PMID 15093881
- [Background] Gassull MA, Cabre E, Vilar L, Alastrue A, Montserrat A. Protein-energy malnutrition: an integral approach and a simple new classification. Hum Nutr Clin Nutr. 1984 Nov;38(6):419-31. PMID 6440876
- [Background] Gastelurrutia P, Lupon J, Domingo M, Ribas N, Noguero M, Martinez C, Cortes M, Bayes-Genis A. Usefulness of body mass index to characterize nutritional status in patients with heart failure. Am J Cardiol. 2011 Oct 15;108(8):1166-70. doi: 10.1016/j.amjcard.2011.06.020. Epub 2011 Jul 26. PMID 21798500